CLINICAL TRIAL: NCT01760954
Title: Extension Study to Evaluate the Long-Term Safety and Efficacy of Elagolix in Subjects With Moderate to Severe Endometriosis-Associated Pain
Brief Title: Study to Evaluate the Long-Term Safety and Efficacy of Elagolix in Adults With Moderate to Severe Endometriosis-Associated Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M12-667
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Results first posted 2018-09-06 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Endometriosis
Keywords: Endometriosis associated pain; Elagolix; Gonadotropin-Releasing Hormone Antagonist; Dysmenorrhea (DYS); Non-Menstrual Pelvic Pain (NMPP)
MeSH Terms: conditions — Endometriosis; Dysmenorrhea | interventions — elagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Elagolix 150 mg QD (Experimental): Participants received elagolix 150 mg tablets once a day (QD) for 6 months.
  Interventions: Drug: Elagolix
- Elagolix 200 mg BID (Experimental): Participants received elagolix 200 mg tablets twice a day (BID) for 6 months.
  Interventions: Drug: Elagolix

INTERVENTIONS:
Drug: Elagolix — Elagolix tablets administered orally
  Other Names: Orilissa™

SUMMARY:
A randomized study evaluating the continued safety and efficacy of elagolix in the management of moderate to severe endometriosis-associated pain in pre-menopausal women.

DETAILED DESCRIPTION:
This is a Phase 3 multicenter, double blind randomized study to assess the continued safety and efficacy of the 150 mg once daily (QD) and 200 mg twice daily (BID) doses of elagolix in premenopausal women with moderate to severe endometriosis-associated pain who completed the 6 month treatment period in the pivotal study M12-665 (NCT01620528). The study consists of 2 periods: a 6 month Treatment Period and a post treatment follow-up period of up to 12 months.

Participants who received elagolix in the pivotal study who met all entry criteria continued to receive the same dose, either elagolix 150 mg QD or elagolix 200 mg BID for up to an additional 6 months in this extension study; participants who received placebo in the pivotal study were randomized in a 1:1 ratio to receive either elagolix 150 mg QD or elagolix 200 mg BID for up to 6 months.

An electronic diary will be used to collect endometriosis-associated pain, uterine bleeding, and analgesic medication use for endometriosis associated pain on a daily basis.

All participants who prematurely discontinued treatment (unless pregnant or elected surgery for endometriosis) or completed the 6-month Treatment Period in this extension study were to enter the Post-treatment Follow-up (PTFU) Period within this study for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Completed the 6 month Treatment Period in pivotal study M12-665 (NCT01620528)
* Agrees to use required birth control methods during the study through Month 6 of the Post-treatment Follow-up period

Exclusion Criteria:

* Clinically significant gynecological condition
* Bone mineral density (BMD) loss greater than or equal to 8 percent in the spine, femoral neck or total hip
* Plans to become pregnant in the next 18 months

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 506 (Actual)
Dates: Start 2012-12-28 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Surrey E, Taylor HS, Giudice L, Lessey BA, Abrao MS, Archer DF, Diamond MP, Johnson NP, Watts NB, Gallagher JC, Simon JA, Carr BR, Dmowski WP, Leyland N, Singh SS, Rechberger T, Agarwal SK, Duan WR, Schwefel B, Thomas JW, Peloso PM, Ng J, Soliman AM, Chwalisz K. Long-Term Outcomes of Elagolix in Women With Endometriosis: Results From Two Extension Studies. Obstet Gynecol. 2018 Jul;132(1):147-160. doi: 10.1097/AOG.0000000000002675. PMID 29889764
- [Derived] Beck D, Winzenborg I, Liu M, Degner J, Mostafa NM, Noertersheuser P, Shebley M. Population Pharmacokinetics of Elagolix in Combination with Low-Dose Estradiol/Norethindrone Acetate in Women with Uterine Fibroids. Clin Pharmacokinet. 2022 Apr;61(4):577-587. doi: 10.1007/s40262-021-01096-w. Epub 2021 Dec 8. PMID 34878624
- [Derived] Stodtmann S, Nader A, Polepally AR, Suleiman AA, Winzenborg I, Noertersheuser P, Ng J, Mostafa NM, Shebley M. Validation of a quantitative systems pharmacology model of calcium homeostasis using elagolix Phase 3 clinical trial data in women with endometriosis. Clin Transl Sci. 2021 Jul;14(4):1611-1619. doi: 10.1111/cts.13040. Epub 2021 May 7. PMID 33963686
- [Derived] Abbas Suleiman A, Nader A, Winzenborg I, Beck D, Polepally AR, Ng J, Noertersheuser P, Mostafa NM. Exposure-Safety Analyses Identify Predictors of Change in Bone Mineral Density and Support Elagolix Labeling for Endometriosis-Associated Pain. CPT Pharmacometrics Syst Pharmacol. 2020 Nov;9(11):639-648. doi: 10.1002/psp4.12560. Epub 2020 Oct 8. PMID 32945631
- [Derived] Winzenborg I, Polepally AR, Nader A, Mostafa NM, Noertersheuser P, Ng J. Effect of Elagolix Exposure on Clinical Efficacy End Points in Phase III Trials in Women With Endometriosis-Associated Pain: An Application of Markov Model. CPT Pharmacometrics Syst Pharmacol. 2020 Aug;9(8):466-475. doi: 10.1002/psp4.12545. Epub 2020 Jul 31. PMID 32621325
- [Derived] Surrey ES, Soliman AM, Agarwal SK, Snabes MC, Diamond MP. Impact of elagolix treatment on fatigue experienced by women with moderate to severe pain associated with endometriosis. Fertil Steril. 2019 Aug;112(2):298-304.e3. doi: 10.1016/j.fertnstert.2019.02.031. Epub 2019 Apr 13. PMID 30992150
- [Derived] Winzenborg I, Nader A, Polepally AR, Liu M, Degner J, Klein CE, Mostafa NM, Noertersheuser P, Ng J. Population Pharmacokinetics of Elagolix in Healthy Women and Women with Endometriosis. Clin Pharmacokinet. 2018 Oct;57(10):1295-1306. doi: 10.1007/s40262-018-0629-6. PMID 29476499

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed the 6-month Treatment Period in the pivotal Study M12-665 (NCT01620528) were eligible to enter this extension study.
  A total of 506 participants were enrolled at 131 sites in the United States, Puerto Rico, and Canada. Two enrolled participants did not receive study drug and are not included in the tables reported below.
Pre-assignment Details: The study consisted of a 6-month Treatment Period and a Post-treatment Follow-up (PTFU) of up to 12 months. Participants who received elagolix in the pivotal study continued to receive the same dose for a further 6 months; participants on placebo in the pivotal study were randomized 1:1 to either elagolix 150 mg once daily or 200 mg twice daily.
Groups:
- Elagolix/Elagolix 150 mg QD: Participants were randomized to elagolix 150 mg once a day (QD) in pivotal Study M12-665 and continued to receive elagolix 150 mg QD for 6 months in this extension Study M12-667.
- Elagolix/Elagolix 200 mg BID: Participants were randomized to elagolix 200 mg twice a day (BID) in pivotal Study M12-665 and continued to receive elagolix 200 mg BID for 6 months in this extension Study M12-667.
- Placebo/Elagolix 150 mg QD: Participants who received placebo in pivotal Study M12-665 and were randomized to elagolix 150 mg QD for 6 months in this extension Study M12-667.
- Placebo/Elagolix 200 mg BID: Participants who received placebo in pivotal Study M12-665 and were randomized to elagolix 200 mg BID for 6 months in this extension Study M12-667.
Period: Treatment Period (6 Months)
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Started | 149 | 138 | 108 | 109
Completed | 116 | 110 | 87 | 83
Not Completed | 33 | 28 | 21 | 26
Not completed — Withdrawal by Subject | 8 | 8 | 4 | 5
Not completed — Adverse Event | 5 | 3 | 4 | 10
Not completed — Lost to Follow-up | 9 | 1 | 4 | 3
Not completed — Surgery or invasive intervention for end | 3 | 3 | 3 | 2
Not completed — Pregnancy | 5 | 0 | 3 | 2
Not completed — Non-compliance | 1 | 4 | 0 | 3
Not completed — Other | 0 | 3 | 3 | 1
Not completed — Decrease in Bone Mineral Density (BMD) | 1 | 6 | 0 | 0
Not completed — Exclusionary Medication | 1 | 0 | 0 | 0
Period: Post-treatment Follow-up (12 Months)
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Started (Participants who completed the 6-month Treatment Period or prematurely discontinued could enter PTFU) | 126 | 118 | 86 | 87
Completed | 96 | 83 | 65 | 67
Not Completed | 30 | 35 | 21 | 20
Not completed — Withdrawal by Subject | 6 | 6 | 4 | 9
Not completed — Lost to Follow-up | 4 | 7 | 2 | 0
Not completed — Surgery or invasive intervention | 6 | 10 | 5 | 5
Not completed — Received Exclusionary Medication | 1 | 4 | 0 | 0
Not completed — Return of Menses and Acceptable BMD | 0 | 0 | 1 | 0
Not completed — Other | 13 | 8 | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID | Total
Number analyzed (Participants) | 149 | 138 | 108 | 109 | 504
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (6.52) | 31.3 (6.32) | 32.4 (6.08) | 32.2 (6.38) | 31.9 (6.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 138 | 108 | 109 | 504
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 21 | 19 | 22 | 85
  Not Hispanic or Latino | 126 | 117 | 89 | 87 | 419
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 133 | 126 | 96 | 95 | 450
  Black or African American | 12 | 9 | 8 | 12 | 41
  Asian | 2 | 0 | 0 | 0 | 2
  American Indian/Alaska Native | 1 | 0 | 1 | 0 | 2
  Multi race | 1 | 3 | 3 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Response for Dysmenorrhea at Month 6 Based on Daily Assessment
Description: Response was defined as a reduction of -0.81 or more from baseline in dysmenorrhea (pain during menstruation) as well as no increase in rescue analgesic use for endometriosis-associated pain (defined as a < 15% increase in average rescue analgesic pill count and no additional analgesic). The response threshold represents a clinically meaningful response that was determined in pivotal Study M12-665.
  Participants recorded rescue analgesic use for endometriosis-associated pain daily and dysmenorrhea and its impact on daily activities each day of their period in an electronic diary (e-Diary). Dysmenorrhea was assessed according to the following:
  * 0: No discomfort
  * 1: Mild discomfort but I was easily able to do the things I usually do
  * 2: Moderate discomfort or pain that made it difficult to do some of the things I usually do
  * 3: Severe pain that made it difficult to do the things I usually do.
  Analgesic use and pain scores were averaged over the 35 days prior to each visit.
Time Frame: Baseline (defined as baseline of Study M12-665 for participants who received elagolix in the pivotal study and baseline of the extension study M12-667 for participants who received placebo in the pivotal study) and Month 6
Population: Participants who received at least 1 dose of double-blind study drug in this extension study with available baseline and month 6 data.
Measure: Number; unit: percentage of participants
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Number analyzed (Participants) | 117 | 110 | 86 | 87
percentage of participants | 52.1 | 78.2 | 32.6 | 64.4

2. Primary Outcome: Percentage of Participants With a Response for Non-menstrual Pelvic Pain at Month 6 Based on Daily Assessment
Description: Response was defined as a reduction of -0.36 or greater from baseline for non-menstrual pelvic pain as well as no increase in rescue analgesic use for endometriosis-associated pain (defined as a < 15% increase in average pill count of rescue analgesics and no additional analgesics). The response threshold represents a clinically meaningful response that was determined in pivotal Study M12-665.
  Participants recorded rescue analgesic medication for endometriosis-associated pain and assessed non-menstrual pelvic pain and its impact on their daily activities each day in an e-Diary according to the following response options:
  * 0: No discomfort
  * 1: Mild discomfort but I was easily able to do the things I usually do
  * 2: Moderate discomfort or pain that made it difficult to do some of the things I usually do
  * 3: Severe pain that made it difficult to do the things I usually do.
  Pain scores and analgesic use were averaged over the 35 days prior to each visit.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Number analyzed (Participants) | 117 | 110 | 86 | 87
percentage of participants | 67.5 | 69.1 | 39.5 | 57.5

3. Secondary Outcome: Percentage of Participants With a Response for Dysmenorrhea at Each Month Based on Daily Assessment
Description: Response was defined as a reduction of -0.81 or more from baseline in dysmenorrhea as well as no increase in rescue analgesic use for endometriosis-associated pain (defined as a < 15% increase in average pill count of rescue analgesics and no additional analgesic). The response threshold represents a clinically meaningful response that was determined in pivotal Study M12-665.
  Participants recorded rescue analgesic medication for endometriosis-associated pain daily and dysmenorrhea (pain during menstruation) and its impact on their daily activities each day of their period in an e-Diary. Dysmenorrhea was assessed according to the following:
  * 0: No discomfort
  * 1: Mild discomfort but I was easily able to do the things I usually do
  * 2: Moderate discomfort or pain that made it difficult to do some of the things I usually do
  * 3: Severe pain that made it difficult to do the things I usually do.
  Analgesic use and pain scores were averaged over the 35 days prior to each visit.
Time Frame: Baseline (defined as baseline of Study M12-665 for participants who received elagolix in the pivotal study and baseline of the extension study M12-667 for participants who received placebo in the pivotal study) and months 1, 2, 3, 4, and 5
Population: Participants who received at least 1 dose of double-blind study drug in this extension study and with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Number analyzed (Participants) | 149 | 138 | 108 | 109
percentage of participants
  Month 1: number analyzed (Participants) | 148 | 136 | 105 | 107
  Month 1 | 48.0 | 80.9 | 21.0 | 20.6
  Month 2: number analyzed (Participants) | 139 | 128 | 97 | 100
  Month 2 | 51.1 | 78.9 | 40.2 | 60.0
  Month 3: number analyzed (Participants) | 132 | 123 | 95 | 94
  Month 3 | 49.2 | 80.5 | 36.8 | 54.3
  Month 4: number analyzed (Participants) | 128 | 119 | 91 | 91
  Month 4 | 53.9 | 79.8 | 39.6 | 58.2
  Month 5: number analyzed (Participants) | 124 | 114 | 89 | 89
  Month 5 | 54.0 | 83.3 | 32.6 | 64.0

4. Secondary Outcome: Percentage of Participants With a Response for Non-menstrual Pelvic Pain at Each Month Based on Daily Assessment
Description: as for outcome 2
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Number analyzed (Participants) | 149 | 138 | 108 | 109
percentage of participants
  Month 1: number analyzed (Participants) | 148 | 136 | 105 | 107
  Month 1 | 55.4 | 74.3 | 23.8 | 29.0
  Month 2: number analyzed (Participants) | 139 | 128 | 97 | 100
  Month 2 | 62.6 | 69.5 | 38.1 | 41.0
  Month 3: number analyzed (Participants) | 132 | 123 | 95 | 94
  Month 3 | 61.4 | 70.7 | 33.7 | 45.7
  Month 4: number analyzed (Participants) | 128 | 119 | 91 | 91
  Month 4 | 64.1 | 75.6 | 39.6 | 47.3
  Month 5: number analyzed (Participants) | 124 | 114 | 89 | 89
  Month 5 | 61.3 | 71.9 | 40.4 | 51.7

5. Secondary Outcome: Percentage of Participants With a Response for Dyspareunia at Each Month Based on Daily Assessment
Description: Response was defined as a reduction of -0.36 or more from baseline in dyspareunia (pain during sexual intercourse) as well as no increase in rescue analgesic use for endometriosis-associated pain (defined as a < 15% increase in average rescue analgesic pill count and no additional analgesics).
  Participants recorded rescue analgesic medication for endometriosis-associated pain and assessed dyspareunia each day in an e-Diary. Dyspareunia was assessed according to the following:
  * 0: None; No discomfort during sexual intercourse
  * 1: Mild; Able to tolerate the discomfort during sexual intercourse
  * 2: Moderate; Intercourse was interrupted due to pain
  * 3: Severe; Avoided intercourse because of pain
  * Not applicable; I was not sexually active for reasons other than endometriosis or did not have sexual intercourse.
  Pain scores and analgesic use were averaged over the 35 days prior to each visit. Responses of "Not Applicable" were excluded.
Time Frame: Baseline (defined as baseline of Study M12-665 for participants who received elagolix in the pivotal study and baseline of the extension study M12-667 for participants who received placebo in the pivotal study) and months 1, 2, 3, 4, 5, and 6
Population: Participants who received at least 1 dose of double-blind study drug in this extension study and with available data at each time point; if a participant's mean score was not defined because all reports in that month were "Not Applicable," then that mean score was treated as missing.
Measure: Number; unit: percentage of participants
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Number analyzed (Participants) | 149 | 138 | 108 | 109
percentage of participants
  Month 1: number analyzed (Participants) | 106 | 93 | 72 | 77
  Month 1 | 50.0 | 61.3 | 33.3 | 15.6
  Month 2: number analyzed (Participants) | 104 | 84 | 67 | 70
  Month 2 | 51.9 | 58.3 | 35.8 | 30.0
  Month 3: number analyzed (Participants) | 98 | 80 | 66 | 64
  Month 3 | 50.0 | 63.8 | 36.4 | 32.8
  Month 4: number analyzed (Participants) | 92 | 75 | 64 | 62
  Month 4 | 48.9 | 65.3 | 46.9 | 41.9
  Month 5: number analyzed (Participants) | 88 | 75 | 63 | 58
  Month 5 | 46.6 | 65.3 | 38.1 | 39.7
  Month 6: number analyzed (Participants) | 84 | 70 | 59 | 58
  Month 6 | 45.2 | 60.0 | 39.0 | 43.1

6. Secondary Outcome: Percent Change From Baseline in Dysmenorrhea Based on Daily Assessment
Description: Participants assessed dysmenorrhea (pain during menstruation) and its impact on their daily activities each day of their period in an e-Diary according to the following response options:
  * 0: No discomfort
  * 1: Mild discomfort but I was easily able to do the things I usually do
  * 2: Moderate discomfort or pain that made it difficult to do some of the things I usually do
  * 3: Severe pain that made it difficult to do the things I usually do.
  Pain scores were averaged over the 35 days prior to each visit.
Time Frame: as for outcome 5
Population: Participants who received at least 1 dose of double-blind study drug in this extension study with available baseline data and data at each time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Number analyzed (Participants) | 149 | 138 | 107 | 107
percent change
  Month 1: number analyzed (Participants) | 148 | 136 | 96 | 101
  Month 1 | -46.7 (44.00) | -82.7 (34.81) | -19.0 (50.35) | -19.3 (51.09)
  Month 2: number analyzed (Participants) | 139 | 128 | 89 | 95
  Month 2 | -46.7 (44.93) | -84.8 (29.81) | -46.6 (47.39) | -67.3 (47.74)
  Month 3: number analyzed (Participants) | 132 | 123 | 88 | 89
  Month 3 | -47.9 (42.37) | -84.5 (33.24) | -36.3 (57.28) | -65.9 (47.17)
  Month 4: number analyzed (Participants) | 128 | 119 | 85 | 87
  Month 4 | -51.4 (44.65) | -85.1 (30.52) | -38.2 (52.48) | -67.4 (47.80)
  Month 5: number analyzed (Participants) | 124 | 114 | 84 | 85
  Month 5 | -52.4 (43.55) | -83.4 (31.19) | -33.4 (48.29) | -77.2 (41.90)
  Month 6: number analyzed (Participants) | 117 | 110 | 81 | 83
  Month 6 | -49.2 (43.75) | -82.0 (33.29) | -37.9 (47.43) | -71.6 (47.81)

7. Secondary Outcome: Percent Change From Baseline in Non-menstrual Pelvic Pain Based on Daily Assessment
Description: Participants assessed non-menstrual pelvic pain and its impact on their daily activities each day in an e-Diary according to the following response options:
  * 0: No discomfort
  * 1: Mild discomfort but I was easily able to do the things I usually do
  * 2: Moderate discomfort or pain that made it difficult to do some of the things I usually do
  * 3: Severe pain that made it difficult to do the things I usually do.
  Pain scores were averaged over the 35 days prior to each visit.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Number analyzed (Participants) | 149 | 138 | 107 | 107
percent change
  Month 1: number analyzed (Participants) | 148 | 136 | 103 | 104
  Month 1 | -37.4 (43.90) | -54.5 (40.35) | -9.6 (104.61) | -20.7 (51.24)
  Month 2: number analyzed (Participants) | 139 | 128 | 96 | 97
  Month 2 | -41.4 (41.49) | -56.4 (38.54) | -22.6 (85.60) | -18.0 (98.73)
  Month 3: number analyzed (Participants) | 132 | 123 | 94 | 91
  Month 3 | -44.0 (40.44) | -56.8 (39.14) | -19.7 (93.18) | -30.2 (57.07)
  Month 4: number analyzed (Participants) | 128 | 119 | 90 | 89
  Month 4 | -47.2 (41.30) | -59.6 (37.30) | -32.0 (66.23) | -33.9 (53.27)
  Month 5: number analyzed (Participants) | 124 | 114 | 89 | 87
  Month 5 | -45.3 (41.05) | -58.0 (39.18) | -17.7 (126.45) | -42.5 (43.01)
  Month 6: number analyzed (Participants) | 117 | 110 | 86 | 85
  Month 6 | -48.9 (41.69) | -56.5 (40.15) | -10.2 (163.42) | -43.9 (43.57)

8. Secondary Outcome: Percent Change From Baseline in Dyspareunia Based on Daily Assessment
Description: Participants assessed dyspareunia each day in an e-Diary according to the following response options:
  * 0: None; No discomfort during sexual intercourse
  * 1: Mild; Able to tolerate the discomfort during sexual intercourse
  * 2: Moderate; Intercourse was interrupted due to pain
  * 3: Severe; Avoided intercourse because of pain
  * Not applicable; I was not sexually active for reasons other than endometriosis or did not have sexual intercourse.
  Pain scores were averaged over the 35 days prior to each visit. Responses of "Not Applicable" were excluded.
Time Frame: as for outcome 5
Population: Participants who received at least 1 dose of double-blind study drug in this extension study and with available baseline data and data at each time point; participants with responses of 'Not Applicable' on all reported days during baseline or for the entire time point were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Number analyzed (Participants) | 123 | 109 | 85 | 82
percent change
  Month 1: number analyzed (Participants) | 98 | 89 | 66 | 72
  Month 1 | -32.8 (63.13) | -39.5 (71.30) | -12.9 (62.92) | -1.1 (63.74)
  Month 2: number analyzed (Participants) | 98 | 80 | 61 | 66
  Month 2 | -36.2 (56.97) | -40.4 (63.27) | -16.2 (82.49) | -27.1 (48.17)
  Month 3: number analyzed (Participants) | 93 | 77 | 60 | 60
  Month 3 | -36.1 (55.41) | -38.6 (75.34) | -14.1 (76.54) | -23.5 (50.71)
  Month 4: number analyzed (Participants) | 86 | 72 | 58 | 58
  Month 4 | -35.0 (55.27) | -48.6 (63.81) | -24.3 (76.26) | -20.7 (71.89)
  Month 5: number analyzed (Participants) | 83 | 72 | 57 | 55
  Month 5 | -34.9 (58.90) | -44.8 (76.01) | -20.2 (62.92) | -27.5 (58.78)
  Month 6: number analyzed (Participants) | 79 | 69 | 53 | 56
  Month 6 | -30.7 (66.57) | -41.7 (68.50) | -28.0 (66.59) | -12.6 (107.83)

9. Secondary Outcome: Change From Baseline in Any Rescue Analgesic Use
Description: Permitted rescue analgesics varied by country and were limited to non-steroidal anti-inflammatory drugs (NSAID) (naproxen 500 mg), or opioid analgesics (hydrocodone 5 mg + acetaminophen 300 mg or 325 mg, and/or codeine 30 mg + acetaminophen 300 mg). Use of rescue analgesic medications taken for endometriosis-associated pain was recorded by the participant daily in the e-Diary as the total number of pills/tablets of each type taken within a 24-hour period. Any rescue analgesic use (NSAID and/or opioid) was calculated as the total number of pills divided by the number of days in the window (i.e. average daily pill count) over the 35-day window prior to and including the reference study day.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pills/day
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Number analyzed (Participants) | 149 | 138 | 107 | 107
pills/day
  Month 1: number analyzed (Participants) | 148 | 136 | 105 | 107
  Month 1 | -0.35 (0.743) | -0.58 (0.687) | -0.15 (0.398) | -0.16 (0.486)
  Month 2: number analyzed (Participants) | 139 | 128 | 97 | 100
  Month 2 | -0.35 (0.646) | -0.59 (0.735) | -0.24 (0.471) | -0.28 (0.481)
  Month 3: number analyzed (Participants) | 132 | 123 | 95 | 94
  Month 3 | -0.37 (0.733) | -0.61 (0.785) | -0.25 (0.525) | -0.32 (0.470)
  Month 4: number analyzed (Participants) | 128 | 119 | 91 | 91
  Month 4 | -0.40 (0.703) | -0.62 (0.697) | -0.26 (0.521) | -0.35 (0.616)
  Month 5: number analyzed (Participants) | 124 | 114 | 89 | 89
  Month 5 | -0.41 (0.687) | -0.59 (0.685) | -0.27 (0.626) | -0.34 (0.590)
  Month 6: number analyzed (Participants) | 117 | 110 | 86 | 87
  Month 6 | -0.40 (0.699) | -0.56 (0.667) | -0.22 (0.616) | -0.38 (0.602)

10. Secondary Outcome: Change From Baseline in NSAID Rescue Analgesic Use
Description: Permitted rescue analgesics varied by country and were limited to non-steroidal anti-inflammatory drugs (NSAID) (naproxen 500 mg), or opioid analgesics (hydrocodone 5 mg + acetaminophen 300 mg or 325 mg, and/or codeine 30 mg + acetaminophen 300 mg). Use of rescue analgesic medications taken for endometriosis-associated pain was recorded by the participant daily in the e-Diary as the total number of pills/tablets of each type taken within a 24-hour period. NSAID rescue analgesic use was calculated as the total number of NSAID pills divided by the number of days in the window (i.e. average daily pill count) over the 35-day window prior to and including the reference study day.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pills/day
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Number analyzed (Participants) | 149 | 138 | 107 | 107
pills/day
  Month 1: number analyzed (Participants) | 148 | 136 | 105 | 107
  Month 1 | -0.24 (0.484) | -0.34 (0.469) | -0.07 (0.217) | -0.09 (0.314)
  Month 2: number analyzed (Participants) | 139 | 128 | 97 | 100
  Month 2 | -0.24 (0.472) | -0.34 (0.462) | -0.12 (0.302) | -0.14 (0.311)
  Month 3: number analyzed (Participants) | 132 | 123 | 95 | 94
  Month 3 | -0.24 (0.488) | -0.34 (0.460) | -0.12 (0.324) | -0.14 (0.346)
  Month 4: number analyzed (Participants) | 128 | 119 | 91 | 91
  Month 4 | -0.25 (0.461) | -0.35 (0.450) | -0.13 (0.336) | -0.17 (0.397)
  Month 5: number analyzed (Participants) | 124 | 114 | 89 | 89
  Month 5 | -0.27 (0.494) | -0.32 (0.417) | -0.13 (0.378) | -0.17 (0.394)
  Month 6: number analyzed (Participants) | 117 | 110 | 86 | 87
  Month 6 | -0.27 (0.517) | -0.31 (0.430) | -0.12 (0.380) | -0.23 (0.453)

11. Secondary Outcome: Change From Baseline in Opioid Rescue Analgesic Use
Description: Permitted rescue analgesics varied by country and were limited to non-steroidal anti-inflammatory drugs (NSAID) (naproxen 500 mg), or opioid analgesics (hydrocodone 5 mg + acetaminophen 300 mg or 325 mg, and/or codeine 30 mg + acetaminophen 300 mg). Use of rescue analgesic medications taken for endometriosis-associated pain was recorded by the participant daily in the e-Diary as the total number of pills/tablets of each type taken within a 24-hour period. Opioid rescue analgesic use was calculated as the total number of opioid pills divided by the number of days in the window (i.e. average daily pill count) over the 35-day window prior to and including the reference study day.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pills/day
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Number analyzed (Participants) | 149 | 138 | 107 | 107
pills/day
  Month 1: number analyzed (Participants) | 148 | 136 | 105 | 107
  Month 1 | -0.11 (0.547) | -0.24 (0.469) | -0.09 (0.272) | -0.07 (0.329)
  Month 2: number analyzed (Participants) | 139 | 128 | 97 | 100
  Month 2 | -0.11 (0.441) | -0.25 (0.532) | -0.12 (0.267) | -0.14 (0.344)
  Month 3: number analyzed (Participants) | 132 | 123 | 95 | 94
  Month 3 | -0.13 (0.540) | -0.28 (0.599) | -0.13 (0.298) | -0.17 (0.338)
  Month 4: number analyzed (Participants) | 128 | 119 | 91 | 91
  Month 4 | -0.15 (0.541) | -0.27 (0.581) | -0.13 (0.298) | -0.19 (0.501)
  Month 5: number analyzed (Participants) | 124 | 114 | 89 | 89
  Month 5 | -0.15 (0.469) | -0.27 (0.558) | -0.14 (0.384) | -0.17 (0.444)
  Month 6: number analyzed (Participants) | 117 | 110 | 86 | 87
  Month 6 | -0.13 (0.439) | -0.25 (0.534) | -0.10 (0.369) | -0.16 (0.392)

12. Secondary Outcome: Percent Change From Baseline in Endometriosis-Associated Pain Score Assessed With Numeric Rating Scale (NRS)
Description: The NRS measured endometriosis-associated pain with and without menstruation on an 11-point scale from 0 = no pain to 10 = worst pain ever. Participants were asked to assess their endometriosis pain over the past 24 hours at it's worst at approximately the same time every day in the e-Diary. Pain scores were averaged over the 35 days prior to each visit.
Time Frame: as for outcome 5
Population: Participants who received at least 1 dose of double-blind study drug in this extension study and with available baseline data and data at each time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Number analyzed (Participants) | 149 | 138 | 107 | 107
percent change
  Month 1: number analyzed (Participants) | 148 | 136 | 104 | 107
  Month 1 | -41.0 (39.85) | -60.0 (36.93) | -9.2 (81.63) | -22.3 (34.41)
  Month 2: number analyzed (Participants) | 139 | 128 | 96 | 100
  Month 2 | -44.4 (38.35) | -62.1 (33.80) | -31.2 (39.22) | -34.6 (41.07)
  Month 3: number analyzed (Participants) | 132 | 123 | 94 | 94
  Month 3 | -45.5 (36.23) | -62.2 (34.10) | -28.0 (55.94) | -39.9 (41.48)
  Month 4: number analyzed (Participants) | 128 | 119 | 90 | 91
  Month 4 | -47.7 (37.99) | -63.5 (32.93) | -32.8 (57.74) | -40.0 (54.65)
  Month 5: number analyzed (Participants) | 124 | 114 | 89 | 89
  Month 5 | -46.4 (38.07) | -62.1 (34.56) | -29.0 (71.65) | -46.4 (39.07)
  Month 6: number analyzed (Participants) | 117 | 110 | 86 | 87
  Month 6 | -48.2 (38.97) | -60.7 (36.09) | -27.8 (64.75) | -45.5 (44.10)

13. Secondary Outcome: Percentage of Participants With a PGIC Response of Much Improved or Very Much Improved
Description: The Patient Global Impression of Change (PGIC) is a questionnaire-based assessment of the change in endometriosis pain since the initiation of study drug. The participant was asked to select from one of seven response categories:
  1. Very Much Improved
  2. Much Improved
  3. Minimally Improved
  4. Not Changed
  5. Minimally Worse
  6. Much Worse
  7. Very Much Worse
Time Frame: Months 1, 2, 3, 4, 5, and 6
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Number analyzed (Participants) | 149 | 148 | 108 | 109
percentage of participants
  Month 1: number analyzed (Participants) | 139 | 132 | 102 | 101
  Month 1 | 63.3 | 86.4 | 47.1 | 45.5
  Month 2: number analyzed (Participants) | 136 | 126 | 99 | 100
  Month 2 | 64.7 | 87.3 | 65.7 | 70.0
  Month 3: number analyzed (Participants) | 129 | 119 | 95 | 94
  Month 3 | 64.3 | 87.4 | 73.7 | 71.3
  Month 4: number analyzed (Participants) | 123 | 118 | 92 | 89
  Month 4 | 70.7 | 91.5 | 73.9 | 70.8
  Month 5: number analyzed (Participants) | 121 | 112 | 86 | 89
  Month 5 | 75.2 | 87.5 | 66.3 | 78.7
  Month 6: number analyzed (Participants) | 111 | 102 | 81 | 82
  Month 6 | 69.4 | 91.2 | 70.4 | 79.3

14. Secondary Outcome: Change From Baseline in Endometriosis Health Profile-30 (EHP-30) Pain Dimension
Description: The EHP-30 is an instrument to measure health-related quality of life in women with endometriosis. The EHP-30 consists of two parts: a core questionnaire containing 5 scales that are applicable to all women with endometriosis and includes pain, control and powerlessness, emotional well-being, social support, and self-image, and a modular part containing 6 scales which do not necessarily apply to all women with endometriosis.
  Each question in the core questionnaire is scored on the following scale: 0 = Never, 1 = Rarely, 2 = Sometimes, 3 = Often, 4 = Always.
  The pain dimension consists of 11 questions. The dimension score ranges from 0 to 100, where 0 = best possible health status as measured by the questionnaire; 100 = worst possible health status. A negative change from baseline score indicates improvement in quality of life.
Time Frame: Baseline (defined as baseline of Study M12-665 for participants who received elagolix in the pivotal study and baseline of the extension study M12-667 for participants who received placebo in the pivotal study) and months 1, 3, and 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Number analyzed (Participants) | 149 | 135 | 108 | 109
units on a scale
  Month 1: number analyzed (Participants) | 138 | 127 | 101 | 100
  Month 1 | -29.50 (20.917) | -40.28 (21.503) | -12.98 (17.426) | -13.27 (17.010)
  Month 3: number analyzed (Participants) | 132 | 120 | 94 | 95
  Month 3 | -30.10 (20.231) | -43.16 (20.951) | -17.87 (21.160) | -21.87 (24.087)
  Month 6: number analyzed (Participants) | 107 | 99 | 72 | 80
  Month 6 | -31.18 (22.213) | -41.62 (21.553) | -15.63 (22.676) | -25.17 (23.387)

15. Secondary Outcome: Change From Baseline in Endometriosis Health Profile-30 (EHP-30) Sexual Intercourse Dimension
Description: The EHP-30 is an instrument to measure health-related quality of life in women with endometriosis. The EHP-30 consists of two parts: a core questionnaire containing 5 scales that are applicable to all women with endometriosis and a modular part containing 6 scales which do not necessarily apply to all women with endometriosis; only 1 modular questionnaire (sexual intercourse [5 items]) was used in this study.
  The Sexual Intercourse dimension consists of 5 questions, each answered on the following scale: 0 = Never, 1 = Rarely, 2 = Sometimes, 3 = Often, 4 = Always, or Not Applicable (not scored). The dimension score ranges from 0 to 100, where 0 = best possible health status as measured by the questionnaire; 100 = worst possible health status. A negative change from baseline score indicates improvement in quality of life.
Time Frame: as for outcome 14
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Number analyzed (Participants) | 120 | 102 | 97 | 95
units on a scale
  Month 1: number analyzed (Participants) | 105 | 86 | 73 | 71
  Month 1 | -19.81 (23.828) | -29.42 (28.257) | -8.15 (21.287) | -9.86 (17.484)
  Month 3: number analyzed (Participants) | 97 | 77 | 72 | 68
  Month 3 | -20.88 (24.979) | -27.27 (30.431) | -15.00 (22.890) | -18.24 (23.015)
  Month 6: number analyzed (Participants) | 78 | 64 | 51 | 52
  Month 6 | -24.23 (27.065) | -30.55 (33.831) | -12.45 (26.858) | -23.17 (25.763)

16. Secondary Outcome: Change From Baseline in Health-Related Productivity Questionnaire (HRPQ): Hours of Work Lost in Workplace and Household
Description: The HRPQ consists of 9 questions measuring the impact of endometriosis-associated pain and its treatment on work productivity and daily activities in the home.
  Absenteeism: Number of hours of intended work lost due to illness or treatment. Presenteeism: Number of hours of work where output was impacted by illness or treatments.
  Total hours lost is the sum of hours missed due to absenteeism plus presenteeism.
Time Frame: as for outcome 1
Population: Participants who received at least 1 dose of double-blind study drug in this extension study with available baseline data and data at each time point. Hours lost from workplace were only calculated for participants who were employed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Number analyzed (Participants) | 140 | 135 | 102 | 106
hours
  Absenteeism from workplace: number analyzed (Participants) | 76 | 72 | 48 | 60
  Absenteeism from workplace | -1.84 (5.636) | -3.01 (6.771) | -2.15 (4.258) | -2.78 (4.730)
  Presenteeism from workplace: number analyzed (Participants) | 76 | 69 | 48 | 59
  Presenteeism from workplace | -11.14 (8.484) | -12.45 (10.464) | -8.29 (8.307) | -10.15 (10.724)
  Total hours of work lost from workplace: number analyzed (Participants) | 76 | 72 | 48 | 60
  Total hours of work lost from workplace | -12.98 (9.662) | -15.15 (11.653) | -10.44 (9.422) | -13.03 (11.911)
  Absenteeism from household: number analyzed (Participants) | 90 | 91 | 63 | 70
  Absenteeism from household | -3.10 (7.588) | -3.69 (4.486) | -3.76 (7.457) | -2.80 (4.971)
  Presenteeism from household: number analyzed (Participants) | 90 | 90 | 62 | 70
  Presenteeism from household | -2.72 (6.459) | -2.49 (4.531) | -2.95 (4.793) | -2.72 (4.698)
  Total hours of work lost from household: number analyzed (Participants) | 90 | 91 | 63 | 70
  Total hours of work lost from household | -5.82 (11.356) | -6.15 (7.628) | -6.90 (11.673) | -5.52 (6.934)

17. Secondary Outcome: Number of Participants With Non-study Health Visits During the Treatment Period
Description: The Health Resource Use Questionnaire (HRUQ) was used to collect information on non-study-related health visits that participants had during the study.
Time Frame: 6 months
Population: Participants who received at least 1 dose of double-blind study drug in this extension study
Measure: Count of Participants; unit: Participants
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Number analyzed (Participants) | 149 | 138 | 108 | 109
Participants | 81 | 68 | 59 | 48

18. Secondary Outcome: Number of Days in Hospital During the Treatment Period
Description: The Health Resource Use Questionnaire (HRUQ) was used to collect information on non-study-related health visits that participants had during the study, including physician visits, hospitalizations and types of procedures received.
Time Frame: 6 months
Population: Participants who received at least 1 dose of double-blind study drug in this extension study and who underwent hospitalization
Measure: Median (Full Range); unit: days
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
Number analyzed (Participants) | 7 | 6 | 5 | 4
days | 2.0 [1 to 6] | 1.5 [1 to 4] | 3.0 [2 to 8] | 1.0 [1 to 2]

ADVERSE EVENTS:
Time Frame: From the date of the first dose of study drug in Study M12-667 through up to 30 days after the last dose of study drug (up to 7 months).
Arm/Group | Elagolix/Elagolix 150 mg QD | Elagolix/Elagolix 200 mg BID | Placebo/Elagolix 150 mg QD | Placebo/Elagolix 200 mg BID
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/138 | 0/108 | 0/109
Serious Adverse Events (participants affected / at risk) | 5/149 | 4/138 | 5/108 | 5/109
Other Adverse Events (participants affected / at risk) | 79/149 | 74/138 | 55/108 | 68/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elagolix/Elagolix 150 mg QD (N=149) | Elagolix/Elagolix 200 mg BID (N=138) | Placebo/Elagolix 150 mg QD (N=108) | Placebo/Elagolix 200 mg BID (N=109)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INCARCERATED UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
JOINT INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AFFECTIVE DISORDER (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OVARIAN CYST (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
PREMENSTRUAL DYSPHORIC DISORDER (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABORTION INDUCED (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elagolix/Elagolix 150 mg QD (N=149) | Elagolix/Elagolix 200 mg BID (N=138) | Placebo/Elagolix 150 mg QD (N=108) | Placebo/Elagolix 200 mg BID (N=109)
ABDOMINAL PAIN (Gastrointestinal disorders) | 7 (7) | 8 (9) | 2 (3) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 7 (8) | 10 (12) | 6 (6) | 11 (12)
FATIGUE (General disorders) | 9 (9) | 5 (5) | 3 (3) | 4 (4)
BRONCHITIS (Infections and infestations) | 8 (8) | 7 (7) | 3 (3) | 3 (3)
INFLUENZA (Infections and infestations) | 6 (6) | 6 (7) | 7 (7) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 9 (9) | 9 (11) | 5 (5) | 3 (3)
SINUSITIS (Infections and infestations) | 10 (10) | 10 (11) | 6 (6) | 10 (10)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 16 (18) | 4 (4) | 5 (5) | 5 (5)
URINARY TRACT INFECTION (Infections and infestations) | 17 (23) | 11 (12) | 10 (10) | 8 (9)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 8 (10) | 6 (6) | 6 (7) | 3 (5)
BONE DENSITY DECREASED (Investigations) | 2 (2) | 9 (9) | 2 (2) | 3 (3)
C-REACTIVE PROTEIN INCREASED (Investigations) | 3 (3) | 7 (7) | 3 (4) | 3 (4)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7) | 2 (2) | 4 (5)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 (7) | 10 (11) | 3 (3) | 5 (5)
HEADACHE (Nervous system disorders) | 10 (11) | 8 (11) | 10 (13) | 15 (20)
ANXIETY (Psychiatric disorders) | 5 (5) | 2 (2) | 6 (6) | 3 (4)
DEPRESSION (Psychiatric disorders) | 8 (8) | 4 (4) | 2 (2) | 0 (0)
INSOMNIA (Psychiatric disorders) | 5 (5) | 5 (6) | 1 (1) | 6 (7)
HOT FLUSH (Vascular disorders) | 6 (7) | 8 (8) | 18 (19) | 33 (38)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.